CLINICAL TRIAL: NCT05464186
Title: Effects of Whole vs. Nonfat Milk Consumption on Body Composition in Children: a 1-Year RCT
Brief Title: Effects of Whole vs. Nonfat Milk Consumption on Body Composition in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Cara B Ebbeling, Co-Director, New Balance Foundation Obesity Prevention Center; Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-P00041990
Record Dates: First submitted 2022-06-27; First posted 2022-07-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned for 1 year to receive home delivery of: 1) Whole milk, 3 cups a day or 2) Nonfat milk, 3 cups a day.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole milk (Experimental): 3 cups a day of whole milk for 1 year
  Interventions: Behavioral: Whole milk
- Nonfat milk (Experimental): 3 cups a day of nonfat milk for 1 year
  Interventions: Behavioral: Nonfat milk

INTERVENTIONS:
Behavioral: Whole milk — Weekly home delivery of whole milk, daily text messages, monthly virtual visits
  Arms: Whole milk
Behavioral: Nonfat milk — Weekly home delivery of nonfat milk, daily text messages, monthly virtual visits
  Arms: Nonfat milk

SUMMARY:
This study will evaluate the effects of whole vs. nonfat milk consumption on body composition, cardiometabolic disease risk factors, and dietary quality.

DETAILED DESCRIPTION:
Background The optimal type of milk is a topic of much debate. Several recent observational studies indicate that consuming whole (full-fat), compared to reduced-fat milk, is associated with less weight gain and decreased cardiometabolic disease risk. The observed beneficial effect of consuming whole milk on body weight may be due to its greater satiety value, leading to consumption of fewer calories from other lower quality (e.g., sugary) foods. Mechanistic studies indicate that substitution of carbohydrate with certain saturated fatty acids in milk increases low-density lipoprotein cholesterol (LDL-C). However, this increase has been attributed to large, buoyant particles that are less atherogenic than small, dense particles; is accompanied by an increase in high-density lipoprotein cholesterol (HDL-C); and may not elevate overall risk compared to carbohydrate.

Specific Aims and Hypotheses

* To examine the effects of milk consumption on body composition (Aim #1) and cardiometabolic disease risk factors (Aim #2). Primary Hypothesis. Consuming whole milk will result in less weight gain compared to consuming nonfat milk. Secondary hypothesis. Consuming whole milk will decrease cardiometabolic disease risk compared to consuming nonfat milk.
* To explore the effects of milk consumption on dietary quality (Aim #3). Exploratory hypothesis. Consuming whole milk will improve overall dietary quality by displacing lower quality foods compared to consuming nonfat milk, particularly among children with low baseline dietary quality.
* (Ancillary Study) To evaluate the effects of milk consumption on risk and prevalence of dental caries.

Design Randomized Controlled Trial. Participants (N=200, aged 9 to 12 years, BMI≥75th percentile) will be randomly assigned for 1 year to receive: 1) Whole milk, 3 cups/d or 2) Nonfat milk, 3 cups/d. To promote adherence to the interventions, the investigators will rely on home delivery of milk using methods consistent with previous successful studies.

Study Outcomes The primary outcome is change in fat mass measured by air displacement plethysmography (BodPod) at 3 time points (baseline and 6 and 12 months). To evaluate cardiometabolic disease risk factors, the investigators will obtain a plasma MetaboProfile®(LabCorp) that includes lipoprotein particle sizes and subfraction concentrations, novel measures of insulin-resistant dyslipoproteinemia and inflammation, and a conventional lipid profile. The investigators will also measure blood pressure.

For the Ancillary Study, outcomes include salivary cariogenicity (pH, flow, and buffering capacity); caries prevalence; dietary quality (cariogenic potential); and serum 25-hydroxyvitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 12 years
* BMI ≥75th percentile for sex and age
* Residence in the Greater Boston catchment area

Exclusion Criteria:

* Aversion to nonfat or whole milk
* Physician diagnosis of major medical illness, eating disorder, or milk allergy (lactose intolerance not exclusionary as lactase treated milk can be provided)
* Plans to move away from the Greater Boston catchment area during the study period
* Plans to be away from home for ≥5 weeks during the study period (e.g., extended summer vacation)
* Change in body weight exceeding 10% during prior year
* Recent adherence to a special diet
* Chronic use of any medication or dietary supplement that could affect study outcomes
* Another member of the family (first degree relative) or household participating in the study

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fat mass | Change from start of trial (time of randomization) through end of trial (12 months)
  Primary outcome for the overall study, main outcome for Specific Aim #1, measured by air displacement plethysmography (BodPod)

SECONDARY OUTCOMES:
Lean body mass | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by air displacement plethysmography (BodPod)
Percent body fat | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by air displacement plethysmography (BodPod)
Height | Change from start of trial (time of randomization) through end of trial (12 months)
  Linear growth
Body mass index (BMI) | Change from start of trial (time of randomization) through end of trial (12 months)
  Weight in kg divided by height in meters squared
Leptin | Change from start of trial (time of randomization) through end of trial (12 months)
  "Satiety" hormone, released by fat cells, measured by ELISA assay
Ghrelin | Change from start of trial (time of randomization) through end of trial (12 months)
  "Hunger" hormone, released primarily in the stomach, measured by ELISA assay
Insulin-like growth factor-1 (IGF-1) | Change from start of trial (time of randomization) through end of trial (12 months)
  Indicator of growth hormone action, measured by ELISA assay
Insulin-like growth factor-binding protein 3 (IGF-BP3) | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by ELISA assay
Lipoprotein insulin resistance (LPIR) | Change from start of trial (time of randomization) through end of trial (12 months)
  Main outcome for Specific Aim #2; a 6-component weighted score of triglyceride-rich, high-density, and low-density lipoprotein particle (TRL-P, HDL-P, LDL-P) sizes and subfraction concentrations (sum of large and very large TRL-P, large HDL-P, small LDL-P), measured by nuclear magnetic resonance spectroscopy
Triglyceride-rich lipoprotein particle (TRL-P) size | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
High-density lipoprotein particle (HDL-P) size | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Low-density lipoprotein particle (LDL-P) size | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Sum of large and very large TRL-P concentration | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Large HDL-P concentration | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Small LDL-P concentration | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Large LDL-P concentration | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by nuclear magnetic resonance spectroscopy
Triglycerides (TG) | Change from start of trial (time of randomization) through end of trial (12 months)
  Part of conventional lipid profile
High-density lipoprotein cholesterol (HDL-C) | Change from start of trial (time of randomization) through end of trial (12 months)
  Part of conventional lipid profile
Low-density lipoprotein cholesterol (LDL-C) | Change from start of trial (time of randomization) through end of trial (12 months)
  Part of conventional lipid profile
Glucose | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured enzymatically using hexokinase method
Insulin | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by electrochemiluminescence immunoassay
Insulin resistance | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by homeostasis model assessment (HOMA), using fasting glucose and insulin concentrations
Adiponectin - total and high molecular weight | Change from start of trial (time of randomization) through end of trial (12 months)
  Hormone released from fat cells, promotes insulin sensitivity and helps regulate blood glucose, measured by ELISA assay
Hemoglobin A1c (HgA1c) | Change from start of trial (time of randomization) through end of trial (12 months)
  Marker of blood glucose control, measured using a system based turbidimetric immunoinhibition
High-sensitivity C-reactive protein (hsCRP) | Change from start of trial (time of randomization) through end of trial (12 months)
  Indicator of chronic inflammation, measured by immunoturbidimetric assay
Interleukin-6 (IL-6) | Change from start of trial (time of randomization) through end of trial (12 months)
  Protein which stimulates synthesis of hsCRP, measured by ELISA assay
Fibrinogen | Change from start of trial (time of randomization) through end of trial (12 months)
  Protein involved in blood clotting, measured by immunoturbidimetric assay
Plasminogen activator inhibitor-1 (PAI-1) | Change from start of trial (time of randomization) through end of trial (12 months)
  Protein involved in blood clotting, measured by ELISA assay
Systolic blood pressure | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by auscultation
Diastolic blood pressure | Change from start of trial (time of randomization) through end of trial (12 months)
  Measured by auscultation
Salivary cariogenicity | Change from start of trial (time of randomization) through end of trial (12 months)
  (Ancillary Study) Risk for dental caries (cavities), measured using the GC Dental America Saliva-Check Buffer Kit (pH, flow, and buffering capacity)
Caries prevalence | Difference between start of trial (time of randomization) and end of trial (12 months)
  (Ancillary Study) Assessed by clinical examination and digital radiograph (x-rays)
Serum 25-hydroxyvitamin D [25(OH)D] | Change from start of trial (time of randomization) through end of trial (12 months)
  (Ancillary Study) Measured by a competitive electrochemiluminescence immunoassay

OTHER OUTCOMES:
Pentadecanoic acid (C15:0) | Change from start of trial (time of randomization) through end of trial (12 months)
  Process measure, biomarker of milk fast consumption, fatty acid in red blood cell membranes which comes primarily from milk fat
Heptadecanoic acid (C17:0) | Change from start of trial (time of randomization) through end of trial (12 months)
  Process measure, biomarker of milk fast consumption, fatty acid in red blood cell membranes which comes primarily from milk fat
trans Palmitoleic acid (tC16:1ω-7) | Change from start of trial (time of randomization) through end of trial (12 months)
  Process measure, biomarker of milk fast consumption, fatty acid in red blood cell membranes which comes primarily from milk fat
Alternative Healthy Eating Index (AHEI) | Change from start of trial (time of randomization) through end of trial (12 months)
  Main outcome for Specific Aim #3, calculated using data from 24-hour dietary recalls
Milk intake | Change from start of trial (time of randomization) through end of trial (12 months)
  Process outcome, measured by 24-hour dietary recalls
Nutrient profile | Change from start of trial (time of randomization) through end of trial (12 months)
  Added sugars, saturated fat, fiber, calcium; measured by 24-hour dietary recalls
Food and beverage intake pattern | Change from start of trial (time of randomization) through end of trial (12 months)
  Vegetables, fruits, legumes, and sugar-sweetened beverages; measured by 24-hour dietary recalls
  (Ancillary Study) Frequency of consuming between-meal-sugar-containing foods or beverages and consumption of foods (grams) with a high cariogenic potential, measured by 24-hour dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Cara B Ebbeling, PhD, Principal Investigator — Boston Children's Hospital; David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- New Balance Foundation Obesity Prevention Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified IPD on Open Science Framework.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The Study Protocol will be posted prior to enrollment of the first study participant. The IPD and Analytic Code for each peer reviewed manuscript from the study will be posted at the time of publication.
Access Criteria: The data will be available to any interested party through Open Science Framework.

REFERENCES:
- [Background] Albala C, Ebbeling CB, Cifuentes M, Lera L, Bustos N, Ludwig DS. Effects of replacing the habitual consumption of sugar-sweetened beverages with milk in Chilean children. Am J Clin Nutr. 2008 Sep;88(3):605-11. doi: 10.1093/ajcn/88.3.605. PMID 18779274
- [Background] Ebbeling CB. Confusion at the milk cooler: opportunity to bolster the evidence base for preventive nutrition. Am J Clin Nutr. 2020 Feb 1;111(2):240-241. doi: 10.1093/ajcn/nqz319. No abstract available. PMID 31901161
- [Background] Willett WC, Ludwig DS. Milk and Health. N Engl J Med. 2020 Feb 13;382(7):644-654. doi: 10.1056/NEJMra1903547. No abstract available. PMID 32053300